CLINICAL TRIAL: NCT02127944
Title: Assessment of Ovarian Reserve Tests in Unexplained Infertile Women
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Guven, Assıstant. Professor., Karadeniz Technical University
Other Study IDs: MS1
Record Dates: First submitted 2014-04-15; First posted 2014-05-01 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Infertility; Infertility, Female
MeSH Terms: conditions — Infertility; Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — SERUM SAMPLES OF PATIENTS WILL BE STORED .THE SERUM SAMPLES DO NOT CONTAIN DNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FERTILE GROUP: WOMEN HAVE NO INFERTILITY PROBLEMS AND HAVE AT LEAST ONE CHILD
- UNEXPLAINED INFERTILE GROUP: WOMEN WITH INFERTILITY PROBLEMS,NO HISTORY OF PREGNANCY AND HAVE NO CHILDREN

SUMMARY:
IN UNEXPLAINED INFERTILITY IN WOMEN ,OVARY RESERVE IS BORDERLINE IF ASSESSED USING HIGH-SENSITIVE TESTS.

DETAILED DESCRIPTION:
IN UNEXPLAINED INFERTILITY OVARIAN RESERVE TESTS WERE ASSESSED.

IN THIS STUDY, A COMPARISON IS DONE BETWEEN 35 WOMEN WITH UNEXPLAINED FERTILITY(THE PATIENT) AND 35 WOMEN WHO DON'T HAVE ANY FERTILITY PROBLEMS AND HAVE AT LEAST A CHILD (THE CONTROL GROUP).

THE STUDY PARTICIPANTS SHOULD HAVE THE FOLLOWING CRITERIA

Inclusion Criteria:

LESS THAN 35 YEARS OLD, MARRIED WOMEN SHOULD HAVE REGULAR MENSES SHOULD HAVE AT LEAST A YEAR OF UNPROTECTED SEX. THE HUSBAND'S SPERMOGRAM SHOULD HAVE NO ABNORMALITIES THE SUBJECT SHOULD HAVE A NORMAL HYSTEROSALPHINGOGRAPHY

Exclusion Criteria:

HAVING ANY SYSTEMIC DISEASE. LONG HISTORY OF ANY DRUG USAGE.

FOR THE CONTROL GROUP

Inclusion Criteria:

LESS THAN 35 YEARS OLD, MARRIED WOMEN SHOULD HAVE REGULAR MENSES AT LEAST HAVE A CHILD THE HUSBAND'S SPERMOGRAM SHOULD HAVE NO ABNORMALITIES THE SUBJECT SHOULD HAVE A NORMAL HYSTEROSALPHINGOGRAPHY

Exclusion Criteria:

HAVING ANY SYSTEMIC DISEASE. LONG HISTORY OF ANY DRUG USAGE.

THE STUDY INCLUDES THE FOLLOWING TESTS BEING DONE ON THE PATIENTS:

THE FOLLOWING HORMONES' LEVELS WERE STUDIED:AMH (ANTI-MULLERIAN HORMONE),FSH (FOLLICULAR STIMULATING HORMONE) , E2 (ESTRADIOL) AND INHIBIN B.THE FORMER THREE HORMONE LEVELS SHOULD BE ASSESSED ON THE THIRD DAY OF MENSES IN THE STUDY,TRANSVAGINAL ULTRASONOGRAPHIC OVARIAN VOLUME ,OVARIAN ANTRAL FOLLICULE NUMBER,OVARIAN STROMAL BLOODFLOW AND OVARIAN ARTERIAL RESISTANCE WAS MEASURED USING DOPPLER ULTRASONOGRAM.

ELIGIBILITY:
Inclusion Criteria:

* LESS THAN 35 YEARS OLD,
* MARRIED WOMEN
* SHOULD HAVE REGULAR MENSES
* SHOULD HAVE AT LEAST A YEAR OF UNPROTECTED SEX.

Exclusion Criteria:

* HAVING ANY SYSTEMIC DISEASE.
* LONG HISTORY OF ANY DRUG USAGE.

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: ALL STUDY PARTICIPANTS SHOULD BE LESS THAN 35 YEARS OLD, MARRIED , SHOULD HAVE REGULAR MENSES AND SHOULD HAVE AT LEAST A YEAR OF UNPROTECTED SEX.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
LEVELS OF OVARIAN RESERVE MARKERS IN THE SERUM | ONE DAY
  AMH (ANTI-MULLERIAN HORMONE),FSH (FOLLICLE STIMULATING HORMONE),E2 (ESTRADIOL)AND INHIBIN -B LEVELS WILL BE TESTED

SECONDARY OUTCOMES:
ULTRASONOGRAPHIC ASSESSMENT OF OVARIAN RESERVE MARKERS | ONE DAY
  OVARIAN ANTRAL FOLLICULE COUNT ,OVARIAN VOLUME MEASUREMENT,OVARIAN DOPPLER -ULTRASONOGRAPHIC ASSESSMENT

CONTACTS AND LOCATIONS:
Overall Officials: SULEYMAN GUVEN, Principal Investigator — KARADENIZ TECHNICAL UNIVERSITY -MEDICAL FACULTY
Locations (1):
- Ktu Farabi Hospital, Trabzon, Turkey (Türkiye)